CLINICAL TRIAL: NCT06092190
Title: Impact of Lower Limb Spasticity on Tibial Nerve Entrapment in Patients With Stroke
Brief Title: Effect of Spasticity on Tibial Nerve Entrapment
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: October 6 University (Other)
Responsible Party: Principal Investigator, Hosam Magdy Metwally, Lecturer of physical therapy for neurology, October 6 University
Other Study IDs: 2020
Record Dates: First submitted 2023-10-14; First posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Neuropathy; Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A
  Interventions: Device: EMG
- Group B
  Interventions: Device: EMG

INTERVENTIONS:
Device: EMG — Electrodiagnostic testing (electromyography and nerve conduction velocity) can objectively verify the tibial nerve dysfunction. Electrodiagnosis rests upon demonstrating impaired tibial nerve conduction across the tarsal tunnel in context of normal conduction

SUMMARY:
Stroke is the most common cause of mortality and is one of the most common causes of morbidity in the world. Polyneuropathies and entrapment neuropathies are known as the complications of stroke

ELIGIBILITY:
Inclusion Criteria:

* 1- A hundred patients with hemiplegia /paresis subsequent to a stroke as diagnosed by CT or MRI.

  2- A hundred patients from both sexes, their ages ranged from (55-65) years. 3- Body weight of patients was ranged from(55 -95 kg) ,while their height was from (151-185 cm) and BMI was ranged from (20-30 kg/m2).

  4- Duration of illness (6 - 9 months post stroke). 5- Patients have spasticity ranging from grade 1 to grade 3 according to modified Ashworth scale 6- Patients were medically stable

Exclusion Criteria:

* 1- Patients with lumbosacral sciatica that could mimic TTS or interfere with its evaluation 2- Patients with tibial neuropathy, significant polyneuropathy, or marked orthopedic abnormalities; 3- Patients with contractures 4- Patients with psychological disturbance or seizures 5- Systemic diseases known to cause TTS, such as diabetes mellitus, hypothyroidism, rheumatoid arthritis, or chronic renal failure;

Ages: 55 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A hundred patients were selected from the Out-Patient Clinics of Neurology in Kasr Al- Aini Hospitals and Out-Patient Clinic of Neurology, Faculty of Physical Therapy, Cairo University.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2023-03-20 (Actual); Primary Completion 2023-06-20 (Actual); Study Completion 2023-10-20 (Estimated)

PRIMARY OUTCOMES:
Electrodiagnostic testing | 30 minutes
  Electrodiagnostic testing (electromyography and nerve conduction velocity) can objectively verify the tibial nerve dysfunction. Electrodiagnosis rests upon demonstrating impaired tibial nerve conduction across the tarsal tunnel in context of normal conduction. Compression results in damage to the myelin sheath and manifests as delayed latencies and slowed conduction velocities

CONTACTS AND LOCATIONS:
Overall Officials: Hosam Magdy Metwally Abd Alhamid, Ph.D, Principal Investigator — October 6 University; Ahmed Magdy Alshimy, Ph.D, Principal Investigator — Al Ryada University for science and technology
Locations (1):
- October 6 University, Cairo, Egypt